CLINICAL TRIAL: NCT03867851
Title: Open, Randomized, Active Comparator-controlled, Multi-Center Study to Evaluate Safety and Efficacy of IBsolvMIR® in Islet Transplantation
Brief Title: Study to Evaluate Safety and Efficacy of IBsolvMIR in Islet Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow patient recruitment
Sponsor: TikoMed AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NNCIT-02
Record Dates: First submitted 2019-03-05; First posted 2019-03-08 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBsolvMIR (Experimental): Study drug IBsolvMIR administered intravenously at 18 mg/kg on day of transplantation and 3 mg/kg on post-operative days 1, 3, 6.
  Interventions: Drug: IBsolvMIR
- Heparin (Active Comparator): Heparin treatment according to clinical praxis.
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: IBsolvMIR — Study drug IBsolvMIR
  Arms: IBsolvMIR
Drug: Heparin — Clinical praxis
  Arms: Heparin

SUMMARY:
This is a Phase II open, randomized, active comparator-controlled multi center study in patients with severe type-1 diabetes. This is a two-armed study where patients are randomized in a 2:1 ratio between IBsolvMIR and heparin. Eighteen patients are planned to be included.

The study consists of up to 8 visits; screening, transplantation surgery with bolus administration of study drug or active comparator, IBsolvMIR doses on day 1, 3 and 6 after surgery, follow up visits on day 7 and 14, and follow-up phone call on day 44.

The primary endpoint is to study AEs up to 44 days following study drug administration. The secondary endpoints are to evaluate changes in TAT, C-peptide, C3a and HGF at baseline and during the first 24 hours after study drug administration, as well as evaluate a change in levels of C-peptide-glucose-creatinine ratio on day 14 compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Patient on a waiting list for islet transplantation
2. Male and female patients age 18 to 60 years of age.
3. Ability to understand and provide written informed consent.
4. Mentally stable and able to comply with the procedures of the study protocol.
5. Clinical history compatible with type 1 diabetes with onset of disease at < 40 years of age and insulin-dependence for > 5 years at the time of enrolment.
6. Documented C-peptide <0.1 nmol/L before first islet transplantation (stimulated in response to a MMTT or other confirmatory method).
7. All subjects must have received medical treatment of their diabetes under the guidance from an experienced endocrinologist. If not previously transplanted the patient must also have;
8. At least one episode of severe hypoglycemia in the past 1 year defined as an event with at least one of the following symptoms; memory loss, confusion, uncontrollable behavior, unusual difficulty in awakening, suspected seizure, loss of consciousness, or visual symptoms, in which the subject was unable to treat him/herself and which was associated with either a blood/plasma glucose level < 54 mg/dl [3.0 mmol/L] or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration OR
9. Reduced awareness of hypoglycemia as defined by a Clarke score of 4 or more.

Exclusion Criteria:

1. Patients with prior organ transplants other than a kidney graft and/or islets. A previous pancreas transplant can be accepted if it failed within the first week due to thrombosis and the graft was removed.
2. Patients with body mass index (BMI) > 30.
3. Insulin requirement > 0.7 Unit/kg/day at screening.
4. Consistently abnormal liver function tests (> 1.5 x ULN on two consecutive measurements > 2 weeks apart) at screening.
5. Proliferative untreated diabetic retinopathy
6. Increased risk for thrombosis (ex. homozygous APC-resistance) or bleeding (INR>1.5)
7. Any history of malignancy except for completely resected squamous or basal cell carcinoma of the skin
8. Patients with increased cardiac risk defined as;

   * unstable coronary artery disease requiring hospitalization or revascularization within 6 months prior to baseline visit
   * chronic heart failure which required hospitalization 30 days prior to baseline visit
9. Patients with active infections, unless treatment is not judged necessary by the investigators
10. Patients with serological evidence of infection with HIV, hepatitis B (patients with serology consistent with previous vaccination and a history of vaccination are acceptable) or hepatitis C.
11. Patients with active peptic ulcer disease, symptomatic gallstones or portal hypertension.
12. Patients who are pregnant or breastfeeding, or who intend to become pregnant.
13. Patients of childbearing potential not willing to use adequate double contraception with < 1% failure rate after the screening visit until the last visit.
14. Active alcohol or substance abuse
15. Patients with evidence of high-level sensitization (PRA> 50% with flow cytometry).
16. Patients with psychological conditions that make it unsafe to undergo islet transplantation or which preclude compliance with prescribed therapy
17. HbA1c > IFCC 100 mmol/mol, at screening.
18. Patients with any condition or any circumstance that in the opinion of the investigator would make it unsafe to undergo treatment with IBsolvMIR.
19. Patients participating in or having participated in any other clinical drug studies in the past four weeks.
20. History of bleeding disorders
21. History of severe hypersensitivity
22. Previous known heparin-induced thrombocytopenia (HIT)
23. Patients with severe hepatic or renal impairment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
Bleeding events | Up to 44 days.
  Bleeding events after islet transplantation with total dose of 27 mg/kg BW IBsolvMIR in comparison to active comparator Heparin
Other AEs/SAEs after islet transplantation | Up to 44 days.
  Other AEs/SAEs after islet transplantation with total dose of 27 mg/kg BW IBsolvMIR in comparison to active comparator Heparin

SECONDARY OUTCOMES:
Difference between groups in levels of biomarkers | Within 7 days.
  Difference between groups in levels of biomarkers after transplantation
Change in C-peptide / (glucose x creatinine) ratio (CPGCR) | Within 14 days.
  Change in CPGCR at day 14 compared to baseline.
  CPGCR is calculated by:
  C-peptide (ng/mL) / ( glucose (mg/dL) x creatinine ratio (mg/dL) )

CONTACTS AND LOCATIONS:
Locations (5):
- Leiden University Medical Center, Leiden, South Holland, Netherlands
- Oslo Universitetssykehus HF, Oslo, Norway
- Sweden (3):
  - Sahlgrenska sjukhuset, Gothenburg
  - Karolinska Universitetssjukhuset Huddinge, Stockholm
  - Akademiska sjukhuset, Uppsala

IPD SHARING:
Plan to Share IPD: No